CLINICAL TRIAL: NCT04788173
Title: Assessment Of Lipid Profile In Cirrhotic Patients And Its Relation To The Disease Severity.
Brief Title: Assessment Of Lipid Profile In Cirrhotic Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, manal mostafa kamel, Resident in Tropical Medicine and Gastroenterology Department, Sohag University
Other Study IDs: Soh-Med-21-02-15
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2021-02

CONDITIONS: Cirrhosis
Keywords: cirrhosis, lipid profile
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cirrhosis is defined anatomically as a diffuse process with fibrosis and nodule formation. It is the result of the fibrogenesis that occurs with chronic liver injury.

Lipoproteins are complexes of lipid and proteins that are essential for transport of soluble vitamins Liver cells play a serious task in the regulation of lipid metabolism. The principal location for lipoprotein and cholesterol synthesis is in the liver.

In healthy individuals, a compound equilibrium is preserved between utilization, biosynthesis, and transfer of lipid fractions.

Many diseases that affect the parenchyma can lead to changes in the structure of lipoproteins and transport throughout the blood.

Nevertheless, in cirrhotic patients, the metabolism of lipid is changed such that glycogen stores are significantly diminished, contributing to malnutrition and biolysis.

DETAILED DESCRIPTION:
Cirrhosis is defined anatomically as a diffuse process with fibrosis and nodule formation. It is the result of the fibrogenesis that occurs with chronic liver injury.

Lipoproteins are complexes of lipid and proteins that are essential for transport of soluble vitamins Liver cells play a serious task in the regulation of lipid metabolism. The principal location for lipoprotein and cholesterol synthesis is in the liver.

In healthy individuals, a compound equilibrium is preserved between utilization, biosynthesis, and transfer of lipid fractions.

Many diseases that affect the parenchyma can lead to changes in the structure of lipoproteins and transport throughout the blood.

Nevertheless, in cirrhotic patients, the metabolism of lipid is changed such that glycogen stores are significantly diminished, contributing to malnutrition and biolysis.

The preceding studies have reported that cirrhotic patients have abnormal metabolism of lipids, especially reduction in cholesterol level and hypobetalipoproteinemia.

These alterations develop together with the progression of liver disease and may be considered as a prognostic markers for liver decompensation.

The maneuvers concerned with the decline of lipid particles in patients with cirrhosis are compound and need multiple researches for complete understanding.

Protein microsomal triglyceride (TG) transfer protein -+ MTP], enzymatic (acylCoA: cholesterol acyltransferase), and apoprotein (Apo AI) reduction are considered to be linked to these changes.

Owing to the wide occurrence of liver disease in Egypt, we made this study to assess lipid profile in cirrhotic patients and to evaluate its relation to the degree of cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients .

Exclusion Criteria:

* 1-Patients with diabetes mellitus,malignancy,uremia. 2-Patients with history of drugs for dyslipidemia. 3- Patients presented with hepatocellular carcinoma 4- Wilsons disease. 5-Rheumatoid arthritis. 6- Systemic lupus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis. Diagnosis of liver cirrhosis depend on clinical, laboratory, and radiological finding.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Measurement of the lipid profile in cirrhotic patients and compare its levels with normal persons. | 15 weeks from start point.
  Via measurement the levels of triglyceride (TG), total cholesterol,very low-density lipoprotein, low density lipoprotien (LDH), and high-density lipoprotien (HDL) in cirrhotic patients and compare with the control.

SECONDARY OUTCOMES:
Measurement the degree of liver cirrhosis severity and its relationship to lipid profile levels. | 15 weeks from start point
  Via detecting degree of cirrhosis (according to Child score ) and its relation to the degree of lipid profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided